CLINICAL TRIAL: NCT04414046
Title: Study of TCR Alpha Beta T-Cell and CD19 B-Cell Depletion for Hematopoietic Cell Transplantation From Haploidentical Donors in the Treatment of Primary Immunodeficiency and Inherited Metabolic Disorders in Children
Brief Title: TCR Alpha Beta T-cell Depleted Haploidentical HCT in the Treatment of Primary Immunodeficiency and Inherited Metabolic Disorders in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAP-PID; IRB00249754 (Other: JHU ACH IRB)
Record Dates: First submitted 2020-05-24; First posted 2020-06-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Primary Immune Deficiency Disorders; Metabolic Disease
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TCR alpha beta T cell depletion (Experimental): The leukapheresis product will undergo TCR alpha beta negative selection following a standardized protocol
  Interventions: Biological: Haploidentical Hematopoietic Cell Transplantation

INTERVENTIONS:
Biological: Haploidentical Hematopoietic Cell Transplantation — TCR alpha beta T-cell and CD19 B-cell depleted haploidentical transplantation

SUMMARY:
This research is being done to learn if a new type of haploidentical transplantation using TCR alpha beta and CD19 depleted stem cell graft from the donor is safe and effective to treat the patient's underlying condition. This study will use stem cells obtained via peripheral blood or bone marrow from parent or other half-matched family member donor. These will be processed through a special device called CliniMACS, which is considered investigational.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with any form of primary immune deficiency/dysregulatory disorders characterized by aberrant immune function, abnormal hematopoiesis, systemic or organ specific autoimmunity and/or non-malignant lymphoproliferation. This includes, but not limited to:

   I. Disorders of phagocytes: Chronic granulomatous disease, Leukocyte adhesion deficiency, defects of IL-10 pathway, MonoMac syndrome

   II. Defects of cellular and humoral immunity: Severe Combined Immunodeficiency Disorder (infants with classic SCID up to 2 years of age will be excluded due to other open protocol), X-linked hyper-IgM syndrome, DOCK8 deficiency, ZAP70 deficiency, common variable immunodeficiency (CVID), Wiskott-Aldrich syndrome, NEMO deficiency.

   III. Disorder of immune dysregulation: Immunodysregulation polyendocrinopathy enteropathy X-linked (IPEX) syndrome, CTLA4 deficiency, LRBA deficiency, STAT1 GOF, STAT3 GOF, X-linked lymphoproliferative disease etc.

   IV. Other PIDs and immune dysregulatory disorders who can be benefitted by HCT as deemed appropriate by the PI and the treating immunologist.
2. Histiocytic disorders including hemophagocytic lymphohistiocytosis (familial HLH (types 1-5), secondary HLH (refractory to therapy or with recurrent episodes of hyper inflammation) and multisystem refractory Langerhans cell histiocytosis.
3. Metabolic disorders that could improve or stabilize after stem cell transplantation such as mucopolysaccharidoses, neurodegenerative disorders, osteopetrosis, etc.

Inclusion Criteria:

1. Patient has a suitable genotypic identical match of 5/10. The donor and recipient must be identical, as determined by high resolution typing, at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-C, HLA-DRB1 and HLA-DQB1.
2. Patients must have adequate organ function measured by:

   1. Cardiac: asymptomatic or if symptomatic then LVEF at rest must be ≥ 40% or SF ≥ 26%
   2. Pulmonary: asymptomatic or if symptomatic DLCO ≥ 40% of predicted (corrected for hemoglobin) or pulse oximetry ≥ 92% on room air if the patient is unable to perform pulmonary function testing.
   3. Renal: Creatinine clearance (CrCl) or glomerular filtration rate (GFR) must be > 50 mL/min/1.73 m2.
   4. Hepatic: Serum conjugated (direct) bilirubin < 2.0 x ULN for age; AST and ALT < 5.0 x ULN for age.
   5. Karnofsky or Lansky (age-dependent) performance score ≥ 50
3. Signed written informed consent

Exclusion Criteria:

1. Participants who have an HLA-matched sibling who is able and willing to donate bone marrow. Patients with a HLA-matched unrelated donors are not excluded.
2. Pregnant or breastfeeding females.
3. Patient has HIV or uncontrolled fungal, bacterial or viral infections.
4. Patient has received prior solid organ transplant.
5. Patient has active GVHD (> grade II) or chronic extensive GVHD due to a previous allograft at the time of inclusion.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of successful donor engraftment | Day 100 after transplantation
  The incidence of engraftment at day 100 will be described based on donor chimerism in the whole blood and or fractions sorted for T-cell and myeloid subsets. The donor chimerism will be scored as autologous reconstitution (< 5% donor), mixed chimerism (5-49%=low mixed, 50-95%=high mixed), > 95%=full donor chimerism.

SECONDARY OUTCOMES:
Overall survival and Event-free survival | Up to 2 years post transplant
  Overall survival is defined as the time of enrollment to death from any cause or last follow up.
  Event-free survival is defined as the time of enrollment to death, primary or secondary graft failure, graft failure necessitating a second HCT procedure, DLI or stem cell boost given for treatment of falling chimerism, or disease recurrence
Kinetics of neutrophil engraftment | Up to 42 days post transplant
  Neutrophil engraftment defined as absolute neutrophil count ≥500/μL for 3 consecutive measurements on different days
Kinetics of platelet engraftment | Up to 42 days post transplant
  Platelet engraftment defined as sustained platelet count >20,000/μL and >50,000//μL with no platelet transfusions in the preceding seven days.
Transplant-related mortality | Up to 100 days post transplant
  Rate of transplant-related mortality
Acute grade II-IV GvHD | Up to 2 years post transplant
  Incidence and severity of acute graft versus host disease
Chronic GvHD | Up to 2 years post transplant
  Incidence and severity of chronic graft versus host disease
Primary graft failure | Up to 2 years post transplant
  Rates of primary graft failure
Secondary graft failure | Up to 2 years post transplant
  Rates of secondary graft failure
Transplant-related complications | Up to 2 years post transplant
  Frequency of transplant-related complications following transplantation
Transplant-related infections | Up to 2 years post transplant
  Frequency of transplant-related infections following transplantation
Cellular and Immunological reconstitution by laboratory evaluations | Up to 2 years post transplant
  The recovery of different lymphocyte subpopulation (CD3+; CD4+; CD8+; CD3+CD45RA+and CD45RO; TCR alpha beta; TCR gamma delta; CD19+)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Chellapandian, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No